CLINICAL TRIAL: NCT05179005
Title: Zimmer Biomet Patient Outcome and Experience After Chest Wall Repair With RibFix Advantage™
Brief Title: RibFix Advantage™ Post-Market Follow-Up
Acronym: ZB-PIONEER
Status: Terminated | Type: Observational
Why Stopped: Sponsor Terminated
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: 0719-02
Record Dates: First submitted 2021-11-30; First posted 2022-01-05 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Rib Fractures
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- RibFix Advantage: Underwent surgical stabilization of rib fractures
  Interventions: Device: RibFix Advantage

INTERVENTIONS:
Device: RibFix Advantage — Intrathoracic rib fracture stabilization

SUMMARY:
To confirm safety, performance, and clinical benefits for the use of RibFix Advantage™ in the fixation, stabilization, and fusion of rib fractures and osteotomies of normal and osteoporotic bone

DETAILED DESCRIPTION:
Retrospective review of subject demographic and hospital data with a prospective follow-up component evaluating clinical outcomes and quality of life for patients receiving RibFix Advantage for surgical stabilization of rib fractures from 2019 to 2021

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age, male or female
* Underwent reconstruction of the chest wall between February 2019 and September 2021 with RibFix Advantage™ for the fixation, stabilization, or fusion of rib fractures
* Minimum amount of follow-up data available, including one visit post-surgery
* Willing and able to sign an Informed Consent for research
* Willing and able to and complete a post-operative follow-up survey at least 3 months post-surgery

Exclusion Criteria:

* Latent or active infection with positive culture at the time of implantation
* Documented history of metal sensitivity
* Documented psychiatric condition preventing the patient from following post-op care instructions
* Fixation of the first and/or second (true) vertebrosternal rib
* Bilateral rib fractures
* Concurrent surgical procedures (i.e. splenectomy, aortic disruption repair, diaphragm injury repair, etc.) performed during the same hospitalization
* Lung injury (open pneumothorax, tension pneumothorax, hemothorax > 1L, pulmonary contusion requiring mechanical ventilation)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thoracic trauma comprises 20-25% of all traumas worldwide and constitutes the third most common cause of death after abdominal injury and head trauma in polytrauma patients.
  Thoracic trauma directly accounts for approximately 25% of trauma-related mortality and is a contributing factor in another 25% of such cases. The incidence of rib fractures due to trauma has been reported by various studies to range between 7 and 40%.
  There is no standard treatment for rib fractures, though there are several options. Failure to treat rib fracture pain can lead to reduced movement, cough suppression, and secondary infection.
  The conservative option for caring for a rib fracture involves the non-operative management of pain.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of re-operation | 3 months post-op
  Number of subjects who needed surgical re-intervention related to rib fracture repair

SECONDARY OUTCOMES:
Length of stay in hospital | Day 0 (surgery) to Day 7
  Time spent in hospital following surgery

OTHER OUTCOMES:
Overall quality of life | Before surgery and 3 months post-op
  American Chronic Pain Association Quality of Life scale
Respiratory-related quality of life | 3 months post-op
  Chronic Pulmonary Disease Assessment Test

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W Towe, MD, Principal Investigator — UH Seidman Cancer Center
Locations (2):
- United States (2):
  - UCI Health Surgery Services, Orange, California
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tanaka H, Yukioka T, Yamaguti Y, Shimizu S, Goto H, Matsuda H, Shimazaki S. Surgical stabilization of internal pneumatic stabilization? A prospective randomized study of management of severe flail chest patients. J Trauma. 2002 Apr;52(4):727-32; discussion 732. doi: 10.1097/00005373-200204000-00020. PMID 11956391
- [Background] Granetzny A, Abd El-Aal M, Emam E, Shalaby A, Boseila A. Surgical versus conservative treatment of flail chest. Evaluation of the pulmonary status. Interact Cardiovasc Thorac Surg. 2005 Dec;4(6):583-7. doi: 10.1510/icvts.2005.111807. Epub 2005 Sep 15. PMID 17670487
- [Background] Nirula R, Allen B, Layman R, Falimirski ME, Somberg LB. Rib fracture stabilization in patients sustaining blunt chest injury. Am Surg. 2006 Apr;72(4):307-9. doi: 10.1177/000313480607200405. PMID 16676852
- [Background] Campbell N, Conaglen P, Martin K, Antippa P. Surgical stabilization of rib fractures using Inion OTPS wraps--techniques and quality of life follow-up. J Trauma. 2009 Sep;67(3):596-601. doi: 10.1097/TA.0b013e3181ad8cb7. PMID 19741406
- See also: Rib Trauma Solutions — https://zbthoracic.com/rib-fixation/